CLINICAL TRIAL: NCT07397247
Title: Evaluating Response to Tonic Motor Activation (TOMAC) Therapy for Patients With Restless Legs Syndrome and Dopaminergic Augmentation
Brief Title: Tonic Motor Activation (TOMAC) Therapy in Patients With Restless Legs Syndrome and Dopaminergic Augmentation
Acronym: CT-10
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noctrix Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-10
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Restless Legs Syndrome
Keywords: Tonic Motor Activation; TOMAC; Dopaminergic augmentation; Peripheral nerve stimulation; Sleep disorder
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label interventional study in which all enrolled participants receive Tonic Motor Activation (TOMAC) therapy and are followed over a defined treatment period to assess response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- TOMAC Therapy (Experimental): Participants receive Tonic Motor Activation (TOMAC) therapy using noninvasive peroneal nerve stimulation with investigational settings and are followed over a defined treatment period.
  Interventions: Device: Tonic Motor Activation (TOMAC) Device

INTERVENTIONS:
Device: Tonic Motor Activation (TOMAC) Device — Tonic Motor Activation (TOMAC) therapy is delivered using a noninvasive peroneal nerve stimulation device. Participants use the device according to the study protocol over a defined treatment period. The device is used by participants in the home setting according to study instructions.

SUMMARY:
This study evaluates Tonic Motor Activation (TOMAC) therapy in adults with restless legs syndrome and dopaminergic augmentation. Participants use a noninvasive peroneal nerve stimulation device over a defined treatment period to assess symptom response and medication use.

DETAILED DESCRIPTION:
This study includes a 24-week period during which participants use Tonic Motor Activation (TOMAC) therapy delivered by a noninvasive peroneal nerve stimulation device with investigational settings, including the option for extended-duration stimulation.

Participants are prospectively assigned to receive TOMAC therapy according to a predefined, multi-stage study protocol.

The study consists of two phases: an initial 8-week period of stable medication use with device therapy, followed by a 16-week period during which dopamine agonist medication tapering may occur while device therapy continues, as clinically appropriate.

While statistical power calculations indicate that approximately 15 evaluable participants are sufficient for the primary endpoint, up to 50 participants may be enrolled to improve estimate precision and account for attrition.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older when written informed consent is obtained.
* Diagnosis of restless legs syndrome confirmed by IRLSSG criteria.
* Moderate-severe RLS, IRLS ≥15 points at study entry
* Dopaminergic augmentation based on clinician assessment and ASRS (augmentation severity rating scale) ≥5 points at study entry
* Subject agrees to not change the dose or schedule of antidepressants and sleep medications.
* Currently taking stable dose and schedule of dopamine agonist over the 4 weeks prior to enrollment, with average daily dose >= 25mg Levodopa Equivalent Daily Dose (LEDD, https://pdmedcalc.co.uk/calculator).
* Patient reports ≥3 nights per week in the 30d prior to study entry: waking during the sleep period with RLS symptoms that interfered with sleep re-initiation
* RLS sensory symptoms in lower legs and/or feet are equally or more distressing than RLS sensory symptoms in all other anatomical locations.
* The subject possesses the necessary equipment, internet/phone accessibility, and communication ability to complete electronic questionnaires and respond to electronic communications and phone calls from the research staff throughout the in-home portion of the study.
* The subject has signed a valid, IRB-approved informed consent form and can understand the requirements of the study and instructions for device usage.

Exclusion Criteria:

* Baseline ferritin <75 ng/mL or patient is unwilling to consider iron supplementation.
* IV iron supplementation in the 6 months prior to study entry.
* Change to dose of RLS prescription medication(s) in the 4 weeks prior to study entry.
* Medications that are known to exacerbate RLS symptoms, including: Sedative antihistamines, Tri/tetracyclics, MAOIs, SSRIs and SNRIs, Tramadol, Neuroleptics, Antiemetics, or the anticonvulsants Phenytoin or Methsuximid
* Change in medication that is known to affect RLS symptoms in the 4 weeks prior to study entry (e.g. sleep medication, antihistamines, antidepressants).
* Primary sleep disorder other than RLS that significantly interferes with sleep at the time of screening visit (e.g. obstructive sleep apnea with adherent CPAP usage would not be an exclusion but typical sleep onset latency of >60min on nights without RLS symptoms would be an exclusion).
* Irregular sleep schedule: subject reports that bedtime is typically outside of 21:00 - 03:00 or reports that bedtime regularly varies by more than 4 hours, such as due to shift work.
* Subject has neuropathy and is unable to clearly distinguish between symptoms of neuropathy and symptoms of RLS.
* During the initial investigational device titration process, sensation threshold >= 30mA or distraction threshold < 15mA, or the device does not properly fit the subject.
* One or more of the following confounding comorbidities: Stage 4-5 chronic kidney disease or renal failure , Iron-deficient anemia, Severe cardiac disease (NYHA class IV), Movements disorder other than RLS (Parkinson's disease, Huntington's disease, dyskinesia, dystonia), Multiple Sclerosis , Moderate-severe cognitive disorder (MoCA<26) or mental illness, Moderate-severe edema affecting the lower legs
* One or more of the following contraindications to the investigational device: Diagnosis of epilepsy or other seizure disorder, Metal implant in upper fibula, Known allergy to device materials (or severe previous reaction to medical adhesives or bandages), Open sores, or injury at or near the location of therapy device application.
* Known to be pregnant or trying to become pregnant.
* Medical condition not listed above that may affect validity of the study or put the subject at risk as determined by the investigator.
* Subject is using another investigational device or drug during the study.
* Subject does not understand the study requirements or device instructions, does not have the ability to complete the study assessments, or is unable or unwilling to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in IRLS total score at Week 8 relative to Baseline (study entry) | 8 Weeks
  The International Restless Legs Syndrome Study Group (IRLS) Rating Scale is a participant-reported questionnaire assessing the severity of restless legs syndrome symptoms, with total scores ranging from 0 to 40, where higher scores indicate greater severity. The outcome is the change in IRLS total score from baseline (study entry) to Week 8.

SECONDARY OUTCOMES:
Change in MOS-II total score at Week 8 relative to Baseline (study entry) | 8 Weeks
  The Medical Outcomes Study Sleep Problems Index II (MOS-II) score is a subscale of the participant-rated MOS questionnaire that measures subjective sleep quality. The MOS-I (6-items) and MOS-II (9-items) are the two validated subscales of the 12-item MOS Sleep Scale. Both are scored from 0 to 100, where 100 corresponds to the worst possible sleep problems and 0 corresponds to no sleep problems. The mean change is assessed from study entry to Week 8, and the endpoint is evaluated over the past two weeks.
PGI-I responder rate, defined as a PGI-I response of "Very Much Improved" or "Much Improved" at Week 8 | 8 Weeks
  The PGI-I Responder Rate is the percentage of subjects with a Patient Global Impressions of Improvement (PGI-I) rating of Much Improved or Very Much Improved relative to study entry. The scores for the Patient Global Impressions of Improvement (PGI-I) are: Very Much Improved (1), Much Improved (2), Minimally Improved (3), No Change (4), Minimally Worse (5), Much Worse (6), Very Much Worse (7).
  Higher percentage corresponds to better outcome. This outcome will be evaluated at Week 8 relative to study entry.
CGI-I responder rate, defined as a CGI-I response of "Very Much Improved" or "Much Improved" at Week 8 | 8 Weeks
  The CGI-I responder rate is the percentage of subjects with a Clinical Global Impressions of Improvement (CGI-I) rating of Much Improved or Very Much Improved relative to study entry. The scores for the Clinical Global Impressions of Improvement (CGI-I) are: Very Much Improved (1), Much Improved (2), Minimally Improved (3), No Change (4), Minimally Worse (5), Much Worse (6), Very Much Worse (7). Higher percentage corresponds to better outcome. This outcome will be evaluated at Week 8 relative to study entry.
Change in Frequency of RLS symptoms (days/week) at Week 8 relative to Baseline (study entry). | 8 Weeks
  This outcome measures the change in subject-reported number of nights with RLS, derived from a follow up to question 7 of the International Restless Legs Syndrome Study Group (IRLS) questionnaire. The value ranges from 0 to 7 for each time point assessed. The mean change is assessed from study entry to Week 8. A greater decrease represents a better outcome.
Change in Sleep Efficiency percentage at Week 8 compared to baseline (Study entry). | 8 weeks
  Sleep efficiency (SE) is the percentage of the time a person spends asleep relative to the total time dedicated to sleep. A greater increase corresponds to a better outcome.
  During the study, participants will report bedtime, wake-up time, sleep onset latency (SOL), and time awake after sleep onset (WASO) on a daily diary.
  To compute SE percentage: Time in bed (TIB) will be computed as the time between bedtime and wake-up time, Total sleep time (TST) will be computed as (TIB-SOL-WASO), sleep efficiency (SE) percentage will be calculated as 100%*(TST/TIB).
  For each individual participant, the Week 8 data point will correspond to the average of that participant's daily sleep diary responses in Weeks 7 and 8. For each individual participant, the baseline values will be collected at study entry, by asking the participant to recall the average value over the prior 2-week period.
Change in Minutes Awake after Sleep Onset (WASO) at Week 8 relative to baseline (study entry). | 8 Weeks
  Minutes Awake after Sleep Onset (WASO) refer to the total number of minutes awake after first going to sleep and before waking up for the next day in the morning. Greater decrease in WASO corresponds to a better outcome. During the study, participants will report WASO minutes on a daily diary. For each individual participant, the Week 8 data point will correspond to the average of that participant's daily sleep diary responses in Weeks 7 and 8. For each individual participant, the baseline values will be collected at study entry, by asking the participant to recall the average value over the prior 2-week period
Reducer Rate at Week 24 relative to baseline (Study entry). | 24 Weeks
  This outcome assesses the percentage of patients who reduced the Levodopa Equivalent Daily Dose (LEDD) of their RLS medication at Week 24 compared to baseline (study entry).
RLS severity change at Week 24 compared to baseline (study entry). | 24 Weeks
  Change in the International Restless Legs Syndrome Study Group (IRLS) Rating Scale Score, which is a participant rated questionnaire that rates RLS severity from 0-40, where 40 is the most severe. The mean change is assessed from study entry to Week 24.
CGI-I responder rate at Week 24 relative to baseline (study entry) | 24 Weeks
  The CGI-I responder rate is the percentage of subjects with a Clinical Global Impressions of Improvement (CGI-I) rating of Much Improved or Very Much Improved relative to study entry. The scores for the Clinical Global Impressions of Improvement (CGI-I) are: Very Much Improved (1), Much Improved (2), Minimally Improved (3), No Change (4), Minimally Worse (5), Much Worse (6), Very Much Worse (7). Higher percentage corresponds to better outcome.
Change in Levodopa Equivalent Daily Dose (LEDD) at Week 24 compared to baseline (study entry) | 24 Weeks
  Dopaminergic medication doses are converted to levodopa equivalent daily dose (LEDD) using a standardized conversion method. The outcome is the change in LEDD from baseline (study entry) to Week 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared for this study due to the investigational nature of the device and sponsor data governance and confidentiality considerations.